CLINICAL TRIAL: NCT03781817
Title: Intranasal Versus Intravenous Ketamine for Procedural Sedation in Children With Non-operative Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Transition/change of primary investigators
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James Statler, Pediatric Emergency Medicine Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300002731
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Trauma; Fractures, Closed; Children, Only; Deep Sedation; Ketamine
Keywords: procedural sedation; ketamine; pediatric; fracture; intranasal; intravenous; emergency department
MeSH Terms: conditions — Wounds and Injuries; Fractures, Closed; Fractures, Bone; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous ketamine (Active Comparator): Participants randomized to IV ketamine will be receive IV ketamine and Intranasal normal saline.
  Interventions: Drug: Intravenous Ketamine
- Intranasal ketamine (Experimental): Participants randomized to Intranasal Ketamine group will receive Intranasal ketamine and IV normal saline.
  Interventions: Drug: Intranasal Ketamine

INTERVENTIONS:
Drug: Intravenous Ketamine — Subject randomized to IV Ketamine arm will receive IN Normal Saline at induction. After 8 minutes subjects will receive IV Ketamine (10 mg/mL) at a dose of 1.5 mg/kg. Level of sedation will be scored at the 15 minutes from induction to determine if adequate sedation has been achieved.
  Arms: Intravenous ketamine
Drug: Intranasal Ketamine — Subject randomized to IN Ketamine arm will receive IN Ketamine (100 mg/mL) at a dose of 9 mg/kg at induction. After 8 minutes subjects will receive IV Normal Saline. Level of sedation will be scored at the 15 minutes from induction to determine if adequate sedation has been achieved.
  Arms: Intranasal ketamine

SUMMARY:
This a randomized clinical trial involving children with non-operative fractures presenting the emergency department randomized either to intranasal or intravenous ketamine.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Intranasal Ketamine (INK) is efficacious for Procedural Sedation and Analgesia (PSA) when compared to Intravenous Ketamine (IVK) in children with non-operative fractures. The primary aim is to determine if INK provides non-inferior sedation to IVK as defined by a Modified Ramsay Sedation score of ≥ 4 and also to compare the proportion of successful procedure between two treatment groups. The secondary aim is to compare proportion of adverse events and compare duration of sedation and length of emergency department (ED) stay between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-18 years of age.
* American Society of Anesthesiologists (ASA) I or II
* Non-operative fracture requiring reduction
* Body weight less than or equal to 25 kg as measured by standard weighing scale

Exclusion Criteria:

* ASA classification III or above
* Age less than 1 year
* History of hypertension, known coronary artery disease or Kawasaki disease, congestive heart failure, acute glaucoma or globe injury, increased intracranial pressure or intracranial mass lesion, acute porphyria, developmental delays, or major psychiatric disorder
* Prior allergy to ketamine
* Unavailable parent or guardian to provide consent
* Non-English speaking

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Statler, MD, Study Chair — Emory University; Judson Barber, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient screening, enrollment and informed consent will be obtained in the emergency department (ED) of Children's of Alabama (COA). Data collection will take place in the ED as well as in Children's Park Place, Suite 110. The remainder of the research, including data analysis, and collaboration amongst the principal investigator and the sub-investigators, will be conducted in Children's Park Place, Suite 110.
Period: Overall Study
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
Started | 17 | 23
Completed | 17 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Ketamine | Intranasal Ketamine | Total
Number analyzed (Participants) | 17 | 23 | 40
Age, Continuous [Median (Standard Deviation); unit: years] | 5 (1.65) | 5 (1.99) | 5 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 10 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 14 | 19 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Allergies [Count of Participants; unit: Participants] — Whether participants have any previous known medication allergies.
  Participants
    Yes | 0 | 1 | 1
    No | 17 | 22 | 39
Weight (kg) [Mean (Standard Deviation); unit: weight in kilograms] | 18.1 (3.2) | 18.4 (4.13) | 18.15 (3.72)
Past Medical History [Count of Participants; unit: Participants] — Whether participants have any known previous medical history.
  Participants
    Yes | 1 | 4 | 5
    No | 16 | 19 | 35
Past Surgical History [Count of Participants; unit: Participants] — Whether participants have any previous surgical history.
  Participants
    Yes | 1 | 3 | 4
    No | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Adequate Sedation.
Description: Determine if IN ketamine provides non-inferior sedation to IV ketamine as defined by a Modified Ramsay Sedation score of ≥ 4. Modified Ramsay Sedation scale is used to evaluate levels of sedation. The scale range is from 0 to 6 with a higher score indicated deeper levels of sedation. At levels of 4 or greater is set to be satisfactory for deep sedation.
Time Frame: Induction up to 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
Number analyzed (Participants) | 17 | 23
Participants | 17 | 4

2. Primary Outcome: Percentage of Adequately Sedated Participants Successfully Completing the Procedure Without Requiring Rescue Medications.
Description: Rescue medication is defined as requiring additional doses of Ketamine to maintain adequate sedation. Successful procedure completion will be define as completing the procedure with only the induction dose and without requiring rescue medications.
Time Frame: From induction to discharge from sedation by emergency physician, up to 3 hours.
Population: Number of participants that required rescue dosing either due to inadequate sedation at 10 minutes or after adequate sedation at 10 minutes but requiring more sedation to complete the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
Number analyzed (Participants) | 17 | 23
Participants | 7 | 22

3. Secondary Outcome: Percentage of Participants With Non-serious Adverse Events.
Description: Non-serious adverse events include allergic reaction, vomiting, emergence agitation, and oxygen desaturations.
Time Frame: From induction to discharge from the emergency department.
Population: Percentage of participants that experienced any possible adverse events from sedation with either intravenous or intranasal ketamine.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
Number analyzed (Participants) | 17 | 23
Participants
  Yes | 1 | 3
  No | 16 | 20

4. Secondary Outcome: Duration of Sedation Using Modified Ramsay Sedation Scale.
Description: Modified Ramsay Sedation scale is used to evaluate levels of sedation. The scale range is from 0 to 6 with a higher score indicated deeper levels of sedation. At levels of 2 or less is set to be satisfactory for discharge from sedation.
Time Frame: From induction to discharge from sedation by the emergency physician.
Population: Describes the duration of sedation (in minutes) from the start of induction to when participant was discharged from sedation by the emergency physician.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
Number analyzed (Participants) | 17 | 23
Minutes | 65.71 (32.54) | 101.21 (52.4)

5. Secondary Outcome: Duration of Emergency Department Stay.
Description: Measured from time of arrival to emergency department to discharge order.
Time Frame: From arrival to emergency department to discharge order entered by emergency physician.
Population: Duration of total emergency department stay from arrival to the emergency department to discharge order entered by emergency physician.
Measure: Mean (Standard Deviation); unit: Time (in minutes)
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
Number analyzed (Participants) | 17 | 23
Time (in minutes) | 325.65 (104.7) | 312.4 (67.7)

ADVERSE EVENTS:
Time Frame: From the time the induction medication (either intranasal ketamine or intranasal hypertonic saline) to discharge order by the emergency physician, up to 6 hours.
Arm/Group | Intravenous Ketamine | Intranasal Ketamine
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/23
Other Adverse Events (participants affected / at risk) | 1/17 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Ketamine (N=17) | Intranasal Ketamine (N=23)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) — Vomiting after the conclusion of the sedation and procedure not including nausea.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT03781817/Prot_SAP_ICF_002.pdf